CLINICAL TRIAL: NCT04652284
Title: Effectiveness of Rifabutin Triple Therapy for First-line and Rescue Treatment of Helicobacter Pylori Infection
Brief Title: Effectiveness of Rifabutin for Treatment of Helicobacter Pylori
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 900-20-RMC
Record Dates: First submitted 2020-11-01; First posted 2020-12-03 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2020-10

CONDITIONS: Helicobacter Infections; Resistance Bacterial; Gastritis H Pylori
MeSH Terms: conditions — Helicobacter Infections | interventions — Rifabutin; Amoxicillin; Esomeprazole; Clarithromycin; Tinidazole

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, non-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rifabutin full dose (Active Comparator): oral amoxicillin 1000mg bd and rifabutin 150 mg bd and esomeprazole 40 mg bd 14 days
  Interventions: Drug: Rifabutin; Drug: Amoxicillin; Drug: Esomeprazole
- Rifabutin low dose (Active Comparator): oral amoxicillin 1000mg bd and rifabutin 150 mg d and esomeprazole 40 mg bd 14 days
  Interventions: Drug: Rifabutin; Drug: Amoxicillin; Drug: Esomeprazole
- Standard of Care (Active Comparator): Standard of care in previously untreated patients will consist of concomitant treatment (oral amoxicillin 1000mg, clarithromycin 500 mg, tinidazole 500 mg and esomeprazole 40 mg all given twice daily for 14 days). In previously treated patients standard of care will consist of bismuth quadruple therapy, quinolone based therapy, or other susceptibility guided treatment where available
  Interventions: Drug: Amoxicillin; Drug: Esomeprazole; Drug: Clarithromycin; Drug: Tinidazole

INTERVENTIONS:
Drug: Rifabutin — 150 mg
  Other Names: mycobutin®
  Arms: Rifabutin full dose; Rifabutin low dose
Drug: Amoxicillin — 1000 mg
  Other Names: Amoxil®
Drug: Esomeprazole — 40 mg
  Other Names: "nexium"
Drug: Clarithromycin — 500 mg
  Other Names: Biaxin®
  Arms: Standard of Care
Drug: Tinidazole — 500 mg
  Other Names: protocide®
  Arms: Standard of Care

SUMMARY:
The aim of this study is to determine the effectiveness of rifabutin triple therapy for the treatment of H. pylori infection in the Israeli population. Patients with or without a prior history of H. pylori eradication failure will be randomized to receive one of three possible treatments:

Group 1-amoxicillin 1000mg bd and rifabutin 150 mg bd and esomeprazole 40 mg bd Group 2- amoxicillin 1000mg bd and rifabutin 150 mg d and esomeprazole 40 mg bd Group 3- standard of care

DETAILED DESCRIPTION:
Patients who present to the outpatient gastroenterology clinic at our institution with a positive diagnostic test for H pylori will be screened. Included patients will undergo randomisation into 3 groups. Randomization will be performed by a random sequence generator to create equal sized groups in boxes of 12.

Group 1-amoxicillin 1000mg bd and rifabutin 150 mg bd and esomeprazole 40 mg bd Group 2- amoxicillin 1000mg bd and rifabutin 150 mg d and esomeprazole 40 mg bd Group 3- standard of care Standard of care in previously untreated patients will consist of concomitant treatment (amoxicillin 1000mg, clarithromycin 500 mg, tinidazole 500 mg and esomeprazole all given twice daily for 14 days). In previously treated patients standard of care will consist of bismuth quadruple therapy, quinolone based therapy, or other susceptibility guided treatment where available.

Treatment duration will be 14 days in all groups. Patients who are randomised to Group 3 and fail treatment will be offered open label rescue treatment with amoxicillin 1000mg bd, rifabutin 150 mg bd and esomeprazole 40 mg bd (14 days).

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to outpatient clinic with evidence of H. pylori infection

Exclusion Criteria:

* allergy to any of the study drugs
* prior exposure to rifamycin drugs
* inability to provide informed consent
* pregnancy or lactation
* liver disease
* haematological disease
* renal failure
* active malignancy
* immune suppression
* patients not expected to benefit from Helicobacter pylori eradication

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Success of H. pylori treatment | 6 weeks following end of treatment
  Negative 13C-urea breath test or Helicobacter pylori Stool Ag

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | 14 days treatment
  Daily entry of Likert scale (0-10) for the following parameters: diarrhea, nausea, abdominal pain, dyspepsia, reflux, loss of appetite, asthenia and others (free text). Adverse effects leading to treatment discontinuation. Serious adverse events leading to leading to patient's hospitalization, disability, or death, or to birth defects on pregnant patients
Compliance with H. pylori treatment | 14 days treatment
  Assessed by diary entry twice daily. If more than 80% of pills taken, patient considered to be treatment compliant.

CONTACTS AND LOCATIONS:
Overall Officials: Doron Boltin, MBBS, Principal Investigator — Rabin Medical Center

IPD SHARING:
Plan to Share IPD: Yes
anonymized IPD will be available upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: will be available following publication of results for a period of 7 years

REFERENCES:
- [Result] Gingold-Belfer R, Niv Y, Levi Z, Boltin D. Rifabutin triple therapy for first-line and rescue treatment of Helicobacter pylori infection: A systematic review and meta-analysis. J Gastroenterol Hepatol. 2021 Jun;36(6):1392-1402. doi: 10.1111/jgh.15294. Epub 2020 Oct 29. PMID 33037845
- [Result] Graham DY, Canaan Y, Maher J, Wiener G, Hulten KG, Kalfus IN. Rifabutin-Based Triple Therapy (RHB-105) for Helicobacter pylori Eradication: A Double-Blind, Randomized, Controlled Trial. Ann Intern Med. 2020 Jun 16;172(12):795-802. doi: 10.7326/M19-3734. Epub 2020 May 5. PMID 32365359
- [Result] Borody TJ, Pang G, Wettstein AR, Clancy R, Herdman K, Surace R, Llorente R, Ng C. Efficacy and safety of rifabutin-containing 'rescue therapy' for resistant Helicobacter pylori infection. Aliment Pharmacol Ther. 2006 Feb 15;23(4):481-8. doi: 10.1111/j.1365-2036.2006.02793.x. PMID 16441468
- [Result] Perri F, Festa V, Clemente R, Villani MR, Quitadamo M, Caruso N, Bergoli ML, Andriulli A. Randomized study of two "rescue" therapies for Helicobacter pylori-infected patients after failure of standard triple therapies. Am J Gastroenterol. 2001 Jan;96(1):58-62. doi: 10.1111/j.1572-0241.2001.03452.x. PMID 11197288